CLINICAL TRIAL: NCT02725203
Title: Unravelling Effectiveness of a Nurse-led Behavior Change Intervention to Enhance Physical Activity in Patients With a Cardiovascular Risk: a Clustered-randomized Controlled Trial in Primary Care
Brief Title: Unravelling Effectiveness of a Nurse-led Behavior Change Intervention to Enhance Physical Activity in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, H.Westland, RN, MSc, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL54286.041.15
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular risk management; behaviour change techniques; self-management; physical activity; nurse-led; behaviour change wheel; primary care; clustered RCT
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Activate intervention (Experimental): Participants in the intervention arm will visit their primary care nurse four times in a three-month period for structured and comprehensive support in achieving an improved level of physical activity.
  Interventions: Behavioral: Activate
- Control (No Intervention): Patients in the control arm will receive care as usual.

INTERVENTIONS:
Behavioral: Activate — The Activate intervention consists of four nurse-led consultations in a thee-month period. In the consultations patients receive structured and comprehensive support in achieving an improved level of physical activity. The Behavior Change Wheel was used to develop the Activate intervention, and led to a selection of 17 behavior change techniques, which are integrated in the Activate intervention
  Arms: Intervention: Activate intervention

SUMMARY:
A two-armed, cluster randomized controlled trial will be conducted comparing the Activate intervention with care as usual in 31 general practices in the Netherlands, in which approximately 279 patients at risk for cardiovascular disease will participate. The Activate intervention focuses on increasing physical activity and is developed using the Behavior Change Wheel (BCW). The activate intervention consists of four nurse-led consultations divided over a 3-months period. Primary outcome is the level of physical activity measured with an accelerometer. Potential effect modifiers are age, body mass index, level of education, social support, depression, patient-provider relationship and baseline amount of minutes of physical activity. Data will be collected at baseline, at 3 months and at 6 months of follow up.

Nurses will be trained in delivering the intervention by a one-day training and coaching sessions supervised. A process evaluation will be conducted.

DETAILED DESCRIPTION:
Self-management interventions are considered effective in chronic disease patients, but trials have shown inconsistent results and it is unknown which patients benefit most. Adequate self-management requires behaviour change in patients and in healthcare providers to equip them in supporting patients in changing their behaviour. To unravel effectiveness of self-management, a nurse-led intervention was developed targeting at one self-management behaviour, namely physical activity, in primary care patients at risk for cardiovascular disease: the Activate intervention. This study aims to evaluate the effectiveness of the Activate intervention, to identify which patient-related characteristics modify change in physical activity levels in patients at risk for CVD in primary care, and to conduct a process evaluation.

A two-armed, cluster randomized controlled trial will be conducted comparing the Activate intervention with care as usual in 31 general practices in the Netherlands, in which approximately 300 patients at risk for cardiovascular disease will participate. The Activate intervention focuses on increasing physical activity and is developed using the Behavior Change Wheel (BCW). The activate intervention consists of four nurse-led consultations divided over a 3-months period in which 17 behaviour change techniques (BCTs) are integrated. Primary outcome is the level of physical activity measured with an accelerometer . Potential effect modifiers are age, body mass index, level of education, social support, depression, patient-provider relationship and baseline amount of minutes of physical activity. Data will be collected at baseline, at 3 months and at 6 months of follow up.

Subsequently, the BCW was applied to analyse what behavior change is needed in nurses to deliver the Activate intervention adequately. This resulted in a one-day training and coaching sessions supervised by a health psychologist and included 21 BCT.

A process evaluation will be conducted to evaluate the training of nurses, fidelity, dose and reach of the Activate intervention, identify barriers and facilitators for implementation and to assess participants' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Aged 40-75

AND at least one of the following criteria:

* have a high blood pressure (≥ 140 mmHg) or are already treated for high blood pressure
* have a high total cholesterol (≥ 6.5 mmol/l) or already treated for high cholesterol
* have diabetes mellitus type 2 (DM2)
* have a positive family history of CVD AND Do not meet the Dutch Norm for Healthy Exercise according to the Short QUestionnaire to Asses Health (SQUASH).

Exclusion Criteria:

* unable to give informed consent (eg. due to cognitive impairment),
* unable to speak, write and read Dutch,
* have contra-indications to increase their physical activity level (eg. unstable angina pectoris, unstable heart failure, acute illness)
* have a terminal illness or have severe psychiatric illness or chronic disorder(s) that seriously influence the ability to improve their psychical activity level.
* patients should not have participated in a program to increase their level of physical activity in the past 2 years.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
level of physical activity measured with the Personal Activity Monitor (PAM AM300) | baseline - 6 months of follow up
  The amount of minutes of physical activity in the moderate (3-6 METabolic equivalent (METS)) and vigorous categories (≥6 METS) at 6 months of follow up will be considered as primary outcome measure. Patients will be asked to wear the accelerometer during 7 consecutive days for 12 hours a day at baseline (T0), 3 months of follow up (T1) and at 6 months of follow up (T2).

SECONDARY OUTCOMES:
Sedentary behaviour using the accelerometer using amount of minutes in the sedentary category (<1,8 METS) | baseline -3 months and 6 months of follow up
  Sedentary behaviour using the accelerometer using amount of minutes in the sedentary category (<1,8 METS)
Self-efficacy for physical activity using the Exercise Self-efficacy Scale (ESS) | baseline - 3 months and 6 months of follow up
  Self-efficacy for physical activity using the Exercise Self-efficacy Scale (ESS), baseline, T0, T1, T2
Patient activation using the Patient Activation Measure (PAM-13) | baseline -3 months and 6 months of follow up
  Patient activation using the Patient Activation Measure (PAM-13)
Health status using the EQ-5D | baseline - 6 months of follow up
  Health status using the EQ-5D

OTHER OUTCOMES:
Potential effect modifier: age | baseline
  does age modify change in physical activity level
Potential effect modifier: depression using the Hospital Anxiety and Depression Scale (HADS) | baseline
  does depression modify change in physical activity level
Potential effect modifier: Body Mass Index (BMI) | baseline
  does BMI modify change in physical activity level
Potential effect modifier: level of education | baseline
  does education level modify change in physical activity
Potential effect modifier: social support using Multidimensional Scale of Perceived Social Support (MSPSS) | baseline,
  does social support modify change in level of physical activity
Potential effect modifier: patient-provider relationship using the Communication Assessment Tool (CAT) | baseline, 3 months and 6 months of follow up
  does the patient-provider relationship modify change in level of physical activity
Potential effect modifier: baseline amount of minutes of moderate to vigorous level of physical activity using the PAM AM300 | baseline
  does baseline amount of minutes of moderate to vigorous level of physical activity modify change in level of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Marieke J. Schuurmans, PhD, Study Chair — UMC Utrecht; Heleen Westland, MSc, Principal Investigator — UMC Utrecht; Irene D Bos-Touwen, MSc, Principal Investigator — UMC Utrecht; Jaap CA Trappenburg, PhD, Study Chair — UMC Utrecht; Carin D Schröder, PhD, Study Chair — UMC Utrecht
Locations (31):
- Netherlands (31):
  - GP Klaar and Vincent, Ede, Gelderland
  - GP Parklaan, Hoevelaken, Gelderland
  - GP Buren, Buren, Gerlderland
  - GP Emmers, 's-Hertogenbosch, North Brabant
  - GP Lienderweg, Asten, North Brabant
  - GP Timmerman, Drunen, North Brabant
  - GP Tjin a Ton and Parlevliet, Amstelveen, North Holland
  - GP De Kennemerpoort, Bennebroek, North Holland
  - GP Odijk-Visser, Heerhugowaard, North Holland
  - GP Munster, Heerhugowaard, North Holland
  - GP Eedenburgh, Hilversum, North Holland
  - GP Seinhorst, Hilversum, North Holland
  - GP Koedijk, Koedijk, North Holland
  - GP De Hollenhorst, Nieuw-Vennep, North Holland
  - GP Spelt, Wassenaar, North Holland
  - GP Jonker, Colmschate, Overijssel
  - GP Amarant, Kampen, Overijssel
  - GP Rosing and Bruins Slot, Markelo, Overijssel
  - GP Blanker, Thiele, Brand, Zwolle, Overijssel
  - GP Sparreboom, Alphen aan den Rijn, South Holland
  - GP Wiechen, Boskoop, South Holland
  - GP De Wiel, Schoonrewoerd, South Holland
  - GP Mozaiek, The Hague, South Holland
  - GP Loudon, The Hague, South Holland
  - GP Provostlaan, Bilthoven, Utrecht
  - GP van Steenis, Bunnik, Utrecht
  - GP De Bilt, De Bilt, Utrecht
  - GP Tolgaarde, Leusden, Utrecht
  - GP Odijk, Odijk, Utrecht
  - GP De Schans, Woudenberg, Utrecht
  - GP Lombok, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Not yet

REFERENCES:
- [Derived] Westland H, Trappenburg JCA, Schuurmans MJ, Zonneveld MH, Schroder CD. Fidelity of primary care nurses' delivery of a behavioural change intervention enhancing physical activity in patients at risk of cardiovascular disease: an observational study. BMJ Open. 2021 Mar 23;11(3):e046551. doi: 10.1136/bmjopen-2020-046551. PMID 33757957
- [Derived] Westland H, Schuurmans MJ, Bos-Touwen ID, de Bruin-van Leersum MA, Monninkhof EM, Schroder CD, de Vette DA, Trappenburg JC. Effectiveness of the nurse-led Activate intervention in patients at risk of cardiovascular disease in primary care: a cluster-randomised controlled trial. Eur J Cardiovasc Nurs. 2020 Dec;19(8):721-731. doi: 10.1177/1474515120919547. Epub 2020 May 6. PMID 32375491
- [Derived] Westland H, Sluiter J, Te Dorsthorst S, Schroder CD, Trappenburg JCA, Vervoort SCJM, Schuurmans MJ. Patients' experiences with a behaviour change intervention to enhance physical activity in primary care: A mixed methods study. PLoS One. 2019 Feb 12;14(2):e0212169. doi: 10.1371/journal.pone.0212169. eCollection 2019. PMID 30753213
- [Derived] Westland H, Koop Y, Schroder CD, Schuurmans MJ, Slabbers P, Trappenburg JCA, Vervoort SCJM. Nurses' perceptions towards the delivery and feasibility of a behaviour change intervention to enhance physical activity in patients at risk for cardiovascular disease in primary care: a qualitative study. BMC Fam Pract. 2018 Dec 12;19(1):194. doi: 10.1186/s12875-018-0888-1. PMID 30541460
- [Derived] Westland H, Bos-Touwen ID, Trappenburg JC, Schroder CD, de Wit NJ, Schuurmans MJ. Unravelling effectiveness of a nurse-led behaviour change intervention to enhance physical activity in patients at risk for cardiovascular disease in primary care: study protocol for a cluster randomised controlled trial. Trials. 2017 Feb 22;18(1):79. doi: 10.1186/s13063-017-1823-9. PMID 28228151